CLINICAL TRIAL: NCT07190924
Title: The Effect of a CrossFit Training Program on Physical, Physiological, and Hormonal Responses in Untrained Subjects
Brief Title: Inflammatory Responses After CrossFit and Resistance Trainings in Untrained Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Habil Hamdouni (Other)
Responsible Party: Sponsor-Investigator, Habil Hamdouni, Doctor, Institut Supérieur du Sport et de l'Education Physique de Ksar-Saïd
Organization: Institut Supérieur du Sport et de l'Education Physique de Ksar-Saïd (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISS-1386
Record Dates: First submitted 2025-09-14; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Inflammation; Oxidative Stress; Plasma Volume; Hormones
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CrossFit (Experimental): High intensity functional training
  Interventions: Behavioral: 12 week training
- Resistance (Experimental): Periodized resistance training
  Interventions: Behavioral: 12 week training

INTERVENTIONS:
Behavioral: 12 week training — Anti-inflammatory and oxidative environment following 12-weeks of CF training by evaluating inflammatory markers and oxidative precursors in untrained participants
  Arms: CrossFit
Behavioral: 12 week training — Anti-inflammatory and oxidative environment following 12-weeks of resistance training by evaluating inflammatory markers and oxidative precursors in untrained participants
  Arms: Resistance

SUMMARY:
Considering the remarkable increase of the fitness programs, the purpose of this study was to assess and compare the effect of Crossfit (CF) and periodized resistance (RT) trainings on inflammatory/oxidative responses in untrained individuals.

Twenty-four participants (20 men and 4 women, age= 25.7 ± 2.2 years, BMI= 25.7 kg.m-2) were randomly assigned into 12 weeks of these trainings with a rate of five sessions/week. Before and after intervention, participants anthropometric data and graded exercise tests were performed. Before (pre), immediately after (post) and 60min after test (p60) a 20mL venous blood sample were drawn for a later measure of c-reactive protein (CRP), interleukin 1 beta (IL-1ß), tumor necrosis factor alpha (TNF-α), interleukin 6 (IL-6), interleukin 10 (IL-10), thiobarbituric acid reactive substances (TBARS), antioxidant enzymes catalase (CAT) and glutathione peroxidase (GPx).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be non-smokers,
* Participants should not suffer from respiratory issues
* Participants should have healthy kidney and liver
* Participants have no metabolic and neurological disorders

Exclusion Criteria:

* The use of medications during the previous 4 weeks
* Consumption of any product related to anti-inflammatory/oxidative supplements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-04-17 (Actual)

PRIMARY OUTCOMES:
Inflammatory marker | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  c-reactive protein (CRP),
Inflammatory marker | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  interleukin 1 beta (IL-1ß)
Inflammatory marker | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  tumor necrosis factor alpha (TNF-α)
Inflammatory marker | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  interleukin 6 (IL-6)
Inflammatory marker | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  interleukin 10 (IL-10)
Oxidative stress | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  thiobarbituric acid reactive substances (TBARS)
Oxidative stress | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  antioxidant enzymes catalase (CAT)
Oxidative stress | Participants data were performed in one day before beginning the 12 week intervention and one day after the last session
  glutathione peroxidase (GPx)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Supérieur du Sport et de l'Education Physique de Ksar-Saïd, Aryanah, Ariana Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
Under negotation